CLINICAL TRIAL: NCT06478472
Title: Prospective Clinical Study of Orelabrutinib in Combination With Rituximab (OR) for Primary Marginal Zone Lymphoma (MZL) That Failed or Not Suitable for Local Therapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Collaborators: The First Hospital of Jilin University (Other); Fujian Cancer Hospital (Other Government); Guangdong Provincial People's Hospital (Other); Nanfang Hospital, Southern Medical University (Other); The Second Affiliated Hospital of Dalian Medical University (Other); Jiangxi Provincial Cancer Hospital (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Shanxi Provincial Cancer Hospital (Unknown); Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Bing, Xu, Principal Investigator, The First Affiliated Hospital of Xiamen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XMDYYYXYK-09
Record Dates: First submitted 2024-06-23; First posted 2024-06-27 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Marginal Zone Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone | interventions — orelabrutinib; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OR (Experimental): Orelabrutinib in combination with rituximab
  Interventions: Drug: Orelabrutinib in combination with rituximab

INTERVENTIONS:
Drug: Orelabrutinib in combination with rituximab — Induction Phase:
  Orelabrutinib + rituximab for a total of 6 cycles of 28 days each Obrutinib (O) 150mg oral d1-28 Rituximab (R) 375mg/m2 IV d0
  Maintenance phase:
  Orelabrutinib 150mg po qd 24 cycles of 28 days each

SUMMARY:
Orelabrutinib combined with rituximab (OR) therapy were used to assess the efficacy and safety for newly diagnosed Marginal zone cell lymphoma

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≥18 years old, gender is not limited;
2. Histopathologically confirmed CD20-positive marginal zone lymphoma including MALT, SMZL, NMZL;
3. Indications for treatment: impact on organ function, development of symptoms associated with lymphoma, large masses, hematopenia secondary to lymphoma;
4. MZL that has progressed, relapsed, or is unsuitable for local therapy after prior local therapy (local therapy includes surgery, radiotherapy, anti-Helicobacter pylori therapy, anti-hepatitis C therapy);
5. ECOG 0-2;
6. Must have at least one measurable or evaluable lesion using the Lugano 2014 Lymphoma Efficacy Evaluation Criteria: i.e., PET/CT with an evaluable lesion; an intranodal lesion with a long diameter greater than 1.5 cm and a short diameter greater than 1.0 cm or an extranodal lesion with a long diameter of > 1.0 cm, as assessed by CT or MR
7. Participants with splenic MZL who do not meet the above criteria for radiologically measurable disease are eligible, provided that the bone marrow infiltration of the MZL is histologically confirmed;
8. HBV-positive serology (concealed carriers: anti-HBeAg +, HbsAg-, anti-HBsAg +/-) are eligible for enrollment only if they have a negative HBV-DNA test;
9. Major organ function meets the following criteria: a) Blood routine: absolute neutrophil value ≥1.5×109/L, platelet ≥75×109/L, hemoglobin ≥75g/L; if accompanied by bone marrow invasion, absolute neutrophil value ≥1.0×109/L, platelet ≥50×109/L, hemoglobin ≥50g/L; b) Blood biochemistry: total bilirubin ≤1.5 times the ULN, AST or ALT ≤ 2 times ULN; serum creatinine ≤ 1.5 times ULN; serum amylase ≤ ULN; c) Coagulation function: International Normalized Ratio (INR) ≤ 1.5 times ULN. 10) Expected survival ≥ 3 months;
10. Voluntary written informed consent prior to trial screening.

Exclusion Criteria:

1. Lymphoma with CNS involvement or high grade transformation;
2. HIV-positive patients and or HCV-active infection (documented by HCV-RNA-positive test);
3. History of deep vein thrombosis or pulmonary embolism within the last 6 months;
4. Active bleeding within 2 months prior to screening, or taking anticoagulant medications, or in the opinion of the investigator, a definite bleeding tendency
5. Continuous use of drugs with moderate to severe inhibition or strong induction of cytochrome P450 CYP3A;
6. Severe chronic obstructive pulmonary disease (COPD) with hypoxemia.
7. Active bacterial, fungal, or viral infections uncontrolled by systemic therapy;
8. In addition to cured basal cell carcinoma of the skin or cervical cancer in situ or early prostate cancer not requiring systemic therapy, or early breast cancer requiring surgery alone. Other malignant tumors within the last 2 years or concurrently;
9. Uncontrolled or significant cardiovascular disease, including: a) New York Heart Association (NYHA) Class II or higher congestive heart failure, unstable angina, myocardial infarction within 6 months prior to the first dose of study drug, or an arrhythmia requiring treatment with a left ventricular ejection fraction (LVEF) of <50% at the time of Screening; b) primary cardiomyopathies (e.g., dilated cardiomyopathy, hypertrophic cardiomyopathy, hypertrophic cardiomyopathy, cardiomyopathy, cardiomyopathy, cardiomyopathy, cardiomegaly, cardiomyopathy, cardiomegaly) b) Primary cardiomyopathies (e.g., dilated cardiomyopathy, hypertrophic cardiomyopathy, arrhythmogenic right ventricular cardiomyopathy, restrictive cardiomyopathy, indeterminate cardiomyopathy); c) A history of clinically significant prolongation of the QTc interval, or QTc intervals of >470 ms in women and >450 ms in men at Screening; d) Subjects with symptomatic or medically-treated coronary artery heart disease; e) Subjects with difficult-to-control high blood pressure (as determined by a reasonable and tolerable dose of adequate medications based on lifestyle improvement). (blood pressure remains uncontrolled for more than 1 month despite the application of a reasonably tolerable and adequate dose of 3 or more antihypertensive medications (including diuretics) on the basis of lifestyle improvement, or blood pressure is not effectively controlled until 4 or more antihypertensive medications have been administered);
10. Subjects with clinically significant gastrointestinal abnormalities that may interfere with drug ingestion, transit, or absorption (e.g., inability to swallow, chronic diarrhea, intestinal obstruction, etc.), or total gastrectomy;
11. Major surgery within 6 weeks prior to screening or minor surgery within 2 weeks prior to screening. A major surgical procedure is one in which general anesthesia is used, but endoscopy for diagnostic purposes is not considered a major surgical procedure. Insertion of vascular access devices will be exempt from this exclusion criterion; ;
12. Subjects who use drugs or alcohol;
13. Pregnant, lactating females and subjects of childbearing age who do not wish to use contraception;
14. known hypersensitivity or allergic reaction to murine antibodies or proteins
15. Any mental or cognitive impairment that may limit understanding, implementation, and compliance with the informed consent form;
16. Previous treatment with BTK, BCR pathway inhibitors (e.g., PI3K, Syk), and BCL-2 inhibitors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-06-23 (Actual); Primary Completion 2027-06-23 (Estimated); Study Completion 2027-06-23 (Estimated)

PRIMARY OUTCOMES:
CR | Up to 36 months
  Complete remission rate (according to Lugano 2014 criteria)

CONTACTS AND LOCATIONS:
Overall Officials: Bing Xu, Principal Investigator — The First Aiffiliated hosptical of xiamen University
Locations (1):
- Bing, Xu, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: No